CLINICAL TRIAL: NCT01828918
Title: Kaohsiung Medical University Hospital
Brief Title: Biomarkers for the Early Diagnosis, Prediction, Prognosis for Colorectal Cancers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Academia Sinica, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KMUH-IRB-2012-03-02 (II)
Record Dates: First submitted 2013-01-27; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2012-06

CONDITIONS: Colorectal Cancers
Keywords: early diagnosis; prediction; prognosis
MeSH Terms: conditions — Colorectal Neoplasms; Disease | interventions — MicroRNAs

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- early recurrence (Other): find the postoperative early relapse out
  Interventions: Genetic: microRNAs

INTERVENTIONS:
Genetic: microRNAs

SUMMARY:
Recent basic and clinical research on the circulating tumor cells (CTCs) in CRC patients takes potential diagnostics, prognostics, and applications into consideration, especially the molecular detection of CTCs in peripheral blood. Moreover, identification of therapeutic targets on CTCs and real-time monitoring of CTCs in cancer patients undergoing systemic therapy are the most important future clinical applications. CTCs measures may be useful to guide change in treatment decisions.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most frequent malignancies and is also the third major cause of cancer-related death in Taiwan, with over 11,000 new cases of CRC were diagnosed and more than 4,400 Taiwanese died from CRC in 2008 (Department of Health). CRC is regarded as the accumulation of acquired genetic and epigenetic changes causing disorders in cell growth, differentiation and apoptosis resulting in transformation of normal colonic epithelium to colon adenocarcinoma.

Recent basic and clinical research on the circulating tumor cells (CTCs) in CRC patients takes potential diagnostics, prognosis, and applications into consideration, especially the molecular detection of CTCs in peripheral blood. Moreover, identification of therapeutic targets on CTCs and real-time monitoring of CTCs in cancer patients undergoing systemic therapy are the most important future clinical applications. The investigators divide the current project into three dimensions to include all the biomarkers related to diagnostic, prognostic and predictive roles for the potential clinical implication. Sub-project 1: prognostic validation and economic evaluation of biochips/biomarkers. Sub-project 2: evaluation of biomarkers for tailored therapy. Sub-project 3: identification and validation of novel biomarkers for early detection. After accomplishment of three sub-projects, a comprehensive network including early diagnostic, prognostic and predictive biomarkers/biochips for high-risk screening, postoperative surveillance, therapeutic strategies of CRC patients will be formed.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 y/o
2. Histological / pathologic and image study proved colorectal cancer
3. Patients with adequate tissue for biomarkers analysis
4. Patients voluntary sign informed consent

Exclusion Criteria:

* Patients who are not met with either one of items which mentioned above.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
postoperative early recurrence | within 12 months postoperation

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Kaohsiung, Taiwan